CLINICAL TRIAL: NCT00842621
Title: Long Term Effects of Erythrocyte Lysis
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ELYSIS
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Sickle Cell Disease; Hemolytic Anemia
Keywords: Sickle Cell Disease, Hemolytic Anemia; Hemolysis
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia, Hemolytic; Hemolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Serum Plasma Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Pediatric participants with severe sickle cell disease (HbSS or Hb S/β°-thalassemia) who are not receiving treatment, e.g., hydroxyurea or chronic transfusions
  Interventions: Procedure: Clinical Evaluations; Other: Laboratory Studies
- 2: Pediatric participants with other forms of SCD or severe sickle cell disease patients (HbSS or Hb S/β°-thalassemia) being treated with hydroxyurea or chronic transfusions
  Interventions: Procedure: Clinical Evaluations; Other: Laboratory Studies
- 3: Pediatric and adult participants with other non-sickling hematological disorders
  Interventions: Procedure: Clinical Evaluations; Other: Laboratory Studies

INTERVENTIONS:
Procedure: Clinical Evaluations — All clinical evaluations should be performed greater than 30 days from illness or hospitalization. Participants will have weight, height, body mass index (BMI), heart rate, respiratory rate, blood pressure (systolic and diastolic) and pulse oximetry recorded while at rest on room air by clinical staff. Cardiac examination will be performed by echocardiogram.
Other: Laboratory Studies — Blood for:
  Complete Blood Count with Differential, Reticulocyte Count, Micronuclei enumeration, α-globin genotype, G6PD activity, genotype, SNP array,
  Serum for:
  Soluble VCAM-1, ICAM-1, Soluble CD40L, Arginase, Endothelin-1, Prothrombin Fragment 1+2, IL-6, -8, -10, Soluble E-selectin, NOx, Haptoglobin, Tumor necrosis factor alpha
  Plasma for:
  Chemistry 18, Cystatin-C, Ferritin, Lactate Dehydrogenase, C-reactive protein, Erythropoietin, NT-proBNP, Haptoglobin, Von Willibrand Factor Antigen, D-dimer, Factor VIII Assay, Quantitative amino acids, Free hemoglobin, Tumor necrosis factor- α, Thrombin-Antithrombin complex, endothelin-1
  Urine for:
  Urinalysis, Urine spot protein, creatinine, Microalbumin, Urine hemosiderin, Urine hepcidin

SUMMARY:
In this prospective observational trial, participants with chronic hemolysis will be assessed with echocardiogram for elevated tricuspid jet velocity and other evidence of pulmonary hypertension. Participants will have laboratory studies evaluating: severity of hemolysis, splenic function, inflammation, endothelial dysfunction, and hypercoagulability. There will be 3 main categories of participants enrolled in this study: (1) pediatric participants with severe sickle cell disease (SCD) (HbSS, HbS/β° thalassemia ) who are not receiving treatment (e.g., hydroxyurea or chronic transfusions); (2) pediatric participants with other forms of SCD or severe SCD (HbSS, HbS/β° thalassemia) patients being treated with hydroxyurea or chronic transfusions; and (3) pediatric and adult participants with other non-sickling hematological disorders.

DETAILED DESCRIPTION:
1. The study will investigate the relationship between tricuspid regurgitation jet velocity (TRV) and intravascular hemolysis, as measured by serum lactate dehydrogenase (LDH), in untreated children with severe sickle cell disease (HbSS or Hb S/β°-thalassemia)
2. The Study will estimate the prevalence of elevated TRV (≥ 2.5 m/s) in untreated children with severe sickle cell disease (HbSS or Hb S/β°-thalassemia), as measured by echocardiography.

Secondary objectives for this study include the following:

1. To estimate the prevalence of elevated TRV in children with severe sickle cell disease (HbSS or Hb S/β°-thalassemia) receiving hydroxyurea or chronic transfusion therapy.
2. To estimate the prevalence of elevated TRV in children with other forms of hemolytic anemia, including other sickling disorders (such as HbSC or HbS/β+-thalassemia) and non-sickling hemolytic anemia (such as hereditary spherocytosis).
3. To estimate the prevalence of elevated TRV in adults with non-sickling hemolytic anemia, with or without splenic function.
4. To investigate the association between TRV and splenic function
5. To investigate the associations between TRV and laboratory parameters of inflammation and hypercoagulability, such as white blood cell count, platelet count, serum N-terminal pro-brain natriuretic peptide (NT-proBNP),endothelial dysfunction, and other markers of hemolysis (bilirubin, plasma free hemoglobin, haptoglobin, etc.)
6. To evaluate genetic determinants of elevated TRV in children and adults with hemolytic anemia.
7. To investigate changes in TRV and hemolysis over time using serial measurements 2 ± 0.5 years after initial enrollment testing.

ELIGIBILITY:
Inclusion Criteria:

1. Established Diagnosis of Hemolysis

   * Sickle Cell Disease (e.g., HbSS, HbS/β-thalassemia, HbSC)
   * Other conditions with hemolysis (e.g., RBC membranopathies, enzymopathies, unstable hemoglobinopathies, PNH)
2. Age

   * SCD participants: 5 years of age up to 19th birthday
   * All other participants: 5 years of age and up (no age limit)

Exclusion Criteria:

1. Previous cardiac surgery
2. Known left ventricle dysfunction (i.e. shortening fraction < 28%)
3. Known right sided congenital heart defect such as atrial septal defect or pulmonary valve stenosis

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children aged 5 years of age up to 19th birthday with sickle cell disease or other forms of hemolytic anemia; Adults over the age of 18 with non-sickling hemolytic anemia.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2009-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
1.To investigate the relationship between tricuspid regurgitation jet velocity (TRV) and intravascular hemolysis, as measured by serum lactate dehydrogenase (LDH), in untreated children with severe sickle cell disease(HbSS or Hb S/β°-thalassemia. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jane Hankins, MD, MS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Rai P, Okhomina VI, Kang G, Martinez HR, Hankins JS, Joshi V. Longitudinal effect of disease-modifying therapy on left ventricular diastolic function in children with sickle cell anemia. Am J Hematol. 2023 Jun;98(6):838-847. doi: 10.1002/ajh.26911. Epub 2023 Mar 20. PMID 36890729
- [Derived] Whipple NS, Naik RJ, Kang G, Moen J, Govindaswamy SD, Fowler JA, Dowdy J, Penkert R, Joshi VM, Hankins JS. Ventricular global longitudinal strain is altered in children with sickle cell disease. Br J Haematol. 2018 Dec;183(5):796-806. doi: 10.1111/bjh.15607. Epub 2018 Nov 19. PMID 30450553
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols